CLINICAL TRIAL: NCT02879500
Title: Effect of Artificially Sweetened Beverages on Cardiometabolic Risk Factors: A Series of Systematic Reviews and Network Meta-analyses of Randomized Controlled Trials
Brief Title: Network Meta-analyses of Artificially Sweetened Beverages and Cardiometabolic Risk
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: John Sievenpiper (Other)
Responsible Party: Sponsor-Investigator, John Sievenpiper, Associate Professor, University of Toronto
Organization: University of Toronto (Other)
Other Study IDs: DNSG-LCSBs
Record Dates: First submitted 2016-08-22; First posted 2016-08-25 (Estimated); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Overweight; Obesity
Keywords: Systematic review and meta-analysis; Evidence-based medicine (EBM); Evidence-based nutrition (EBN); Clinical practice guidelines; Randomized controlled trials; Prospective cohort studies; Body weight; Body mass index; Adiposity; Overweight; Obesity
MeSH Terms: conditions — Overweight; Obesity; Body Weight | interventions — Artificially Sweetened Beverages

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Diet beverages

SUMMARY:
Sugars especially in form or sugar-sweetened beverages (SSBs) have been singled out as one of the prime culprits in the dual epidemics of obesity and diabetes. Artificially sweetened beverages (ASBs) provide a potentially important means for displacing excess calories from free sugars in the diet. There is, however, a concern that the use of ASBs may themselves contribute to an increased risk of obesity and diabetes. This concern led the 2015 Dietary Guidelines for American Committee (DGAC) to recommend that sugars in the diet not be replaced with ASBs but rather with "healthy options" such as water. Whether ASBs as a replacement strategy for SSBs have the intended benefits and whether these benefits are similar to those of the preferred replacement strategy water remains unclear. To address this important question and update of the European Association of the Study (EASD) clinical practice guidelines for nutrition therapy, the investigators propose to conduct a series of systematic reviews and network meta-analyses of the totality of the evidence from randomized controlled trials to evaluate the effects of water and ASBs on incident overweight and obesity and cardiometabolic risk factors. The findings generated by this proposed knowledge synthesis will help improve the health of consumers through informing evidence/base guidelines and improving health outcomes by educating healthcare providers and patients, stimulating industry innovations, and guiding future research design.

DETAILED DESCRIPTION:
Background: Sugars especially in form or sugar-sweetened beverages (SSBs) have been singled out as one of the prime culprits in the dual epidemics of obesity and diabetes. Artificially sweetened beverages (ASBs) provide a potentially important means for displacing excess calories from free sugars in the diet. There is, however, a concern that the use of ASBs may themselves contribute to an increased risk of obesity and diabetes. This concern led the 2015 Dietary Guidelines for American Committee (DGAC) to recommend that sugars in the diet not be replaced with ASBs but rather with "healthy options" such as water. Whether ASBs as a replacement strategy for SSBs have the intended benefits and whether these benefits are similar to those of the preferred replacement strategy water remains unclear.

Objective: To inform the update of the European Association of the Study (EASD) clinical practice guidelines for nutrition therapy, the investigators will conduct a series of systematic reviews and network meta-analyses to asses the effect of the substitution of ASBs for SSBs, water for SSBs, and ASBs for water on measures of adiposity and cardiometabolic risk factors.

Design: Each systematic review and meta-analysis will be conducted according to the Cochrane Handbook for Systematic Reviews of Interventions and reported according to the Preferred Reporting Items for Systematic Reviews and Meta-Analyses (PRISMA).

Data sources: MEDLINE, EMBASE, and The Cochrane Central Register of Controlled Trials (Clinical Trials; CENTRAL) will be searched using appropriate search terms supplemented by hand searches of references of included studies. Abstracts will be included and no language restrictions will be used.

Study selection: The investigators will include randomized controlled trials (RCTs) that are >=7 days duration and assess the effect of water versus ASBs on incident overweight/obesity or cardiometabolic risk factors.

Data extraction: Two or more investigators will independently extract relevant data and assess risk of bias using the Cochrane Risk of Bias Tool. All disagreements will be resolved by consensus. Standard computations and imputations will be used to derive missing variance data.

Outcomes: There will be 9 outcome clusters. The primary outcome will be body weight. Secondary outcomes will be other markers of adiposity (BMI, body fat, waist circumference); glycemic control (glycated blood proteins [HbA1c, fasting blood glucose, postprandial blood glucose, fasting blood insulin, homeostasis model assessment of insulin resistance [HOMA-IR]); established therapeutic lipid targets (LDL-cholesterol, non-HDL-cholesterol, apolipoprotein B [apo B], HDL-cholesterol, triglycerides, total cholesterol, ); blood pressure (systolic blood pressure and diastolic blood pressure); markers of NAFLD (intrahepatocellular lipids [IHCL], alanine aminotransferase [ALT], aspartate aminotransferase [AST]); and uric acid.

Data synthesis: Risk ratios (incident overweight/obesity) and mean differences (all other outcomes) will be pooled for direct comparisons (ASBs versus water) and indirect comparisons (ASBs versus SSBs and water versus SSBs using SSBs as the common comparator). We will perform Bayesian Network-Meta Analysis (NMA). We will present the pooled estimates as posterior means and 95% credible intervals. We will also use NMA for sensitivity analysis to validate our findings from the conventional generic inverse variance random-effects models. The NMA will be conducted using Markov Chain Monte Carlo (MCMC) approach simulation using GeMTC-R package. Paired analyses will be applied for crossover trials. Heterogeneity will be assessed by the Cochran Q statistic and quantified by the I2 statistic. To explore sources of heterogeneity, the investigators will conduct sensitivity analyses, in which each study is systematically removed. If there are >=10 studies, then the investigators will also explore sources of heterogeneity by a priori subgroup analyses by health status (metabolic syndrome/diabetes, overweight, normal weight), dose (<=median intake, >median intake), baseline measurements (global and abdominal adiposity), randomization, study design (parallel, crossover), energy balance (positive, neutral, negative), follow-up (<=8 weeks, >8 weeks), risk of bias, and individual domains of risk of bias using meta-regression analyses. Meta-regression analyses will assess the significance of categorical and continuous subgroup analyses. When >=10 studies are available, publication bias will be investigated by inspection of funnel plots and formal testing using the Egger test and the Begg test. If publication bias is suspected, then the investigators will attempt to adjust for funnel plot asymmetry by imputing the missing study data using the Duval and Tweedie trim and fill method.

Evidence Assessment: The certainty of the evidence for each outcome will be assessed using the Grading of Recommendations Assessment, Development and Evaluation (GRADE) approach.

Knowledge translation plan: The results will be disseminated through interactive presentations at local, national, and international scientific meetings and publication in high impact factor journals. Target audiences will include the public health and scientific communities with interest in nutrition, diabetes, obesity and cardiovascular disease. Feedback will be incorporated and used to improve the public health message and key areas for future research will be defined. Applicant/Co-applicant decision makers will network among opinion leaders to increase awareness and participate directly as committee members in the development of future guidelines.

Significance: The proposed project will aid in knowledge translation related to the role of ASBs in the development of overweight and obesity, strengthening the evidence-base for guidelines and improving health outcomes by educating healthcare providers and patients, stimulating industry innovation, and guiding future research design.

ELIGIBILITY:
1. RCTs

   Inclusion Criteria:
   * Trials in humans
   * Diet beverage intervention
   * Water comparator
   * Diet duration >= 7 days
   * Viable outcome data

   Exclusion Criteria:
   * Non-human trials
   * Observational studies
   * Lack of suitable comparator
   * Diet duration < 2 weeks
   * No viable outcome data
2. Cohort studies

Inclusion Criteria:

* Prospective cohort studies or case-cohort studies
* Duration >= 1year
* Assessment of the exposure of diet beverages or water
* Ascertainment of viable data by level of exposure

Exclusion Criteria:

* Ecological, cross-sectional, and retrospective observational studies, clinical trials and non-human studies
* Duration < 1 year
* No assessment of exposures of diet beverages or water
* No ascertainment viable clinical outcome data by level of exposure

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All individuals, both children and adults, regardless of health status
Sampling Method: Probability Sample
Enrollment: 1 (Estimated)
Dates: Start 2015-11; Primary Completion 2020-03 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Adiposity - Body weight | Up to 20 years
  body weight

SECONDARY OUTCOMES:
Adiposity - BMI | Up to 20 years
  Body mass index (BMI) in kg/m2
Adiposity - Body fat | Up to 20 years
  Body fat in % (relative units)
Adiposity - waist circumference (WC) | Up to 20 years
  Waist circumference in cm
Glycemic control - HbA1c | Up to 20 years
  HbA1c in % (absolute units)
Glycemic control - fasting plasma glucose (FPG) | Up to 20 years
  Fasting plasma glucose (FPG) in mmol/L
Glycemic control - 2h plasma glucose (2h-PG) | Up to 20 years
  2h plasma glucose (2h-PG) during a 75g oral glucose tolerance test (OGTT) in mmol/L
Glycemic control - fasting plasma insulin (FPI) | Up to 20 years
  Fasting plasma insulin (FPI) in pmol/L
Glycemic control - homeostasis model assessment of insulin resistance (HOMA-IR) | Up to 20 years
  Homeostasis model assessment of insulin resistance (HOMA-IR)
Blood lipid targets - LDL-cholesterol (LDL-C) | Up to 20 years
  LDL-cholesterol (LDL-C) in mmol/L
Blood lipid targets - non-HDL-cholesterol (non-HDL-C) | Up to 20 years
  non-HDL-cholesterol (non-HDL-C) in mmol/L
Blood lipid targets - apolipoprotein B (apo B) | Up to 20 years
  Apolipoprotein B (apo B) in g/L
Blood lipid targets - triglycerides | Up to 20 years
  Triglycerides in mmol/L
Blood lipid targets - HDL-cholesterol (HDL-C) | Up to 20 years
  HDL-cholesterol (HDL-C) in mmol/L
Blood lipid targets - Total-cholesterol (Total-C) | Up to 20 years
  Total-cholesterol (Total-C) in mmol/L
Blood pressure - Systolic blood pressure (SBP) | Up to 20 years
  Systolic blood pressure (SBP) in mmHg
Blood pressure - diastolic blood pressure (DBP) | Up to 20 years
  Diastolic blood pressure (DBP) in mmHg
Markers of non-alcoholic fatty liver disease (NAFLD) - Intrahepatocellular lipids (IHCL) | Up to 20 years
  Intrahepatocellular lipids (IHCL) in % (relative units)
Markers of non-alcoholic fatty liver disease (NAFLD) - alanine transaminase (ALT) | Up to 20 years
  Alanine transaminase (ALT) in U/L
Markers of non-alcoholic fatty liver disease (NAFLD) - aspartate transaminase (AST) | Up to 20 years
  Aspartate transaminase (AST) in U/L
Uric acid | Up to 20 years
  Uric acid in mmol/L

CONTACTS AND LOCATIONS:
Overall Officials: John L Sievenpiper, MD, PhD, FRCPC, Principal Investigator — University of Toronto
Locations (1):
- The Toronto 3D (Diet, Digestive tract and Disease) Knowledge Synthesis and Clinical Trials Unit, Clinical Nutrition and Risk Factor Modification Centre, St. Michael's Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No